CLINICAL TRIAL: NCT07226284
Title: The Effects of Vagus Nerve Stimulation on Intrinsic Lower Leg Spinal Motoneuron Excitability in Parkinson's Disease.
Brief Title: Effects of Vagal Nerve Stimulation on Leg Muscle Activity and Posture in Parkinson's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colum MacKinnon (Other)
Collaborators: Parkinson's Foundation (Other)
Responsible Party: Sponsor-Investigator, Colum MacKinnon, Principal Investigator, University of Minnesota
Organization: University of Minnesota (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NEUR-2025-34303
Record Dates: First submitted 2025-11-03; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: PARKINSON DISEASE (Disorder); Parkinson's Disease (PD)
Keywords: nVNS; Vagus nerve; VNS; Parkinson's disease; PD; gammaCore
MeSH Terms: conditions — Parkinson Disease | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Experiment one will use both a within-subject and cross-sectional design and experiment two will be a double-blind crossover design.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Baseline (no VNS) (Other): Within-subject and cross-sectional design that consists of 30 participants with PD (15 with PIGD and 15 without PIGD) and 15 matched controls.
  Interventions: Other: No intervention
- Real nVNS (Experimental)
  Interventions: Device: Vagal nerve stimulation
- Sham nVNS (Sham Comparator): Sham VNS will be applied using setting that do not active the vagus nerve.
  Interventions: Other: No intervention

INTERVENTIONS:
Device: Vagal nerve stimulation — The gammaCore non-invasive vagus nerve stimulator (nVNS) is a hand-held portable device that is used to apply electrical stimulation to the vagus nerve via two electrodes.
  Arms: Real nVNS
Other: No intervention — No nVNS is applied in the baseline experiment. Sham nVNS is applied for experiment two
  Arms: Baseline (no VNS); Sham nVNS

SUMMARY:
This study is designed to better understand the mechanisms contributing to impaired activation of leg muscles in people with Parkinson's disease (PD) and to test if stimulation of a nerve at the neck can improve muscle activation, walking and balance.

DETAILED DESCRIPTION:
The goals of this project are twofold: (i) to test the hypothesis that persistent inward currents (PICs) in spinal motoneurons of the ankle extensors are reduced in people with Parkinson's disease and that these changes are associated with impaired postural control and (ii) to examine the acute effects of non-invasive vagus nerve stimulation (nVNS) on PICs and postural control.

This project will conduct experiments to test the hypothesis that the firing properties of muscles that control the ankle are significantly altered in people with PD compared to matched healthy adults and that these changes in activity are related to the severity of postural control deficits. In addition, this project will examine the acute effects of non-invasive vagal nerve stimulation (nVNS), an intervention that increases activity in the locus coeruleus and raphe nucleus, on the firing properties of ankle muscles and postural control. If successful, this work will be the first to demonstrate that brainstem pathways that control muscle firing properties are altered in people with PD and are associated with postural impairment. The preliminary trial of nVNS will provide evidence that postural muscle activity can be improved with stimulation and improve postural control. These findings will provide critical preliminary data required to move forward with a clinical trial of nVNS in PD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease,
* On stable medication for the preceding month and anticipated over the next 3 months,
* Able to ambulate without the use of an assistive device for more than 50 meters.

Control Cohort:

* Age (± 3 years) and sex distribution matched to the PD cohort,
* Able to ambulate without the use of an assistive device for more than 50 meters.

Exclusion Criteria:

* Failure to demonstrate capacity to consent (based on UBACC and/or MacArthur-CR),
* History of significant neurological disorder (besides PD in the PD group),
* History of stroke, traumatic brain injury, intracranial aneurysm, intracranial hemorrhage, brain tumor or atypical parkinsonian disorder,
* Severe orthopedic or other related musculoskeletal pathology that has significant adverse effects on gait,
* Women who are pregnant or may be pregnant,
* Insufficient comprehension of the English language,
* History of substance abuse in past 2 years;

Additional exclusion criteria for VNS experiment

* Pain at the nVNS treatment site (e.g., dysesthesia, neuralgia, cervicalgia);
* Lesion (including lymphadenopathy), previous surgery (including carotid endarterectomy or vascular neck surgery) or abnormal anatomy at the stimulation site (open wound, rash, infection, swelling, cut, sore, drug patch, surgical scar[s]);
* Known or suspected severe atherosclerotic cardiovascular disease, severe carotid artery disease (e.g., bruits or history of TIA or stroke), congestive heart failure, known severe coronary artery disease or prior myocardial infarction;
* Abnormal baseline electrocardiogram (ECG) within the last year (e.g., second or third-degree heart block, prolonged QT interval, atrial fibrillation, atrial flutter, history of ventricular tachycardia or ventricular fibrillation);
* Recent history of uncontrolled high blood pressure, bradycardia, tachycardia, or know recent history orthostatic hypotension;
* Previous unilateral or bilateral vagotomy;
* Implanted metal cervical spine hardware, other metallic implants or implantable medical devices such as deep brain stimulator, hearing aid implant, pacemaker, implanted cardioverter defibrillator, cranial aneurysm and/or cranial aneurysm clips, history of facial/orbital/metallic fragments, implanted electronic device, neurostimulator, valve replacements/stents, metallic implants/prostheses) near the stimulation site such as a bone plate or bone screw;
* History of syncope or seizures (within the last 2 years);

Ages: 21 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Change in delta-F | Within-session VNS: 0-60 minutes. Between VNS sessions: 1 - 4 weeks.
  Difference between baseline and post-VNS delta-F measure

SECONDARY OUTCOMES:
Change in Braceheight | Within-session VNS: 0 -60 minutes; between VNS sessions: 1-4 weeks
  Change in brace height measure between before and after VNS
Step length | Within-session VNS: 0-60 minutes; between VNS sessions: 1-4 weeks
  Average step length
Peak magnitude force on step leg | Within-session VNS: 0-60 minutes; between VNS sessions: 1-4 weeks
  peak magnitude of the step leg loading force during gait initiation
Postural sway magnitude | Within-session VNS: 0-60 minutes; between VNS sessions: 1-4 weeks
  Root mean square (RMS) of the center of pressure smoothness (jerk) in the medial-lateral plane.

CONTACTS AND LOCATIONS:
Locations (1):
- Movement Disorders Laboratory, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mondal B, Choudhury S, Simon B, Baker MR, Kumar H. Noninvasive vagus nerve stimulation improves gait and reduces freezing of gait in Parkinson's disease. Mov Disord. 2019 Jun;34(6):917-918. doi: 10.1002/mds.27662. Epub 2019 Mar 14. No abstract available. PMID 30869809
- [Background] Morris R, Yarnall AJ, Hunter H, Taylor JP, Baker MR, Rochester L. Noninvasive vagus nerve stimulation to target gait impairment in Parkinson's disease. Mov Disord. 2019 Jun;34(6):918-919. doi: 10.1002/mds.27664. Epub 2019 Mar 19. No abstract available. PMID 30889295
- [Background] Negro F, Muceli S, Castronovo AM, Holobar A, Farina D. Multi-channel intramuscular and surface EMG decomposition by convolutive blind source separation. J Neural Eng. 2016 Apr;13(2):026027. doi: 10.1088/1741-2560/13/2/026027. Epub 2016 Feb 29. PMID 26924829
- [Background] Stebbins GT, Goetz CG, Burn DJ, Jankovic J, Khoo TK, Tilley BC. How to identify tremor dominant and postural instability/gait difficulty groups with the movement disorder society unified Parkinson's disease rating scale: comparison with the unified Parkinson's disease rating scale. Mov Disord. 2013 May;28(5):668-70. doi: 10.1002/mds.25383. Epub 2013 Feb 13. PMID 23408503
- [Background] Evancho A, Do M, Fortenberry D, Billings R, Sartayev A, Tyler WJ. Vagus nerve stimulation in Parkinson's disease: a scoping review of animal studies and human subjects research. NPJ Parkinsons Dis. 2024 Oct 24;10(1):199. doi: 10.1038/s41531-024-00803-1. PMID 39448636
- [Background] Factor SA, Weinshenker D, McKay JL. A possible pathway to freezing of gait in Parkinson's disease. J Parkinsons Dis. 2025 Mar;15(2):282-290. doi: 10.1177/1877718X241308487. Epub 2025 Jan 14. PMID 39973500
- [Background] Espay AJ, LeWitt PA, Kaufmann H. Norepinephrine deficiency in Parkinson's disease: the case for noradrenergic enhancement. Mov Disord. 2014 Dec;29(14):1710-9. doi: 10.1002/mds.26048. Epub 2014 Oct 9. PMID 25297066
- [Background] Robichaud JA, Pfann KD, Comella CL, Brandabur M, Corcos DM. Greater impairment of extension movements as compared to flexion movements in Parkinson's disease. Exp Brain Res. 2004 May;156(2):240-54. doi: 10.1007/s00221-003-1782-0. Epub 2004 Jan 28. PMID 14747885
- [Background] Pfann KD, Buchman AS, Comella CL, Corcos DM. Control of movement distance in Parkinson's disease. Mov Disord. 2001 Nov;16(6):1048-65. doi: 10.1002/mds.1220. PMID 11748736
- [Background] Folland JP, Haas B, Castle PC. Strength and activation of the knee musculature in Parkinson's disease: effect of medication. NeuroRehabilitation. 2011;29(4):405-11. doi: 10.3233/NRE-2011-0719. PMID 22207069
- [Background] Braak H, Del Tredici K, Rub U, de Vos RA, Jansen Steur EN, Braak E. Staging of brain pathology related to sporadic Parkinson's disease. Neurobiol Aging. 2003 Mar-Apr;24(2):197-211. doi: 10.1016/s0197-4580(02)00065-9. PMID 12498954
- [Background] Kim EH, Wilson JM, Thompson CK, Heckman CJ. Differences in estimated persistent inward currents between ankle flexors and extensors in humans. J Neurophysiol. 2020 Aug 1;124(2):525-535. doi: 10.1152/jn.00746.2019. Epub 2020 Jul 15. PMID 32667263
- [Background] Hulsey DR, Riley JR, Loerwald KW, Rennaker RL 2nd, Kilgard MP, Hays SA. Parametric characterization of neural activity in the locus coeruleus in response to vagus nerve stimulation. Exp Neurol. 2017 Mar;289:21-30. doi: 10.1016/j.expneurol.2016.12.005. Epub 2016 Dec 14. PMID 27988257
- [Background] Gorassini MA, Knash ME, Harvey PJ, Bennett DJ, Yang JF. Role of motoneurons in the generation of muscle spasms after spinal cord injury. Brain. 2004 Oct;127(Pt 10):2247-58. doi: 10.1093/brain/awh243. Epub 2004 Sep 1. PMID 15342360
- [Background] Johnson MD, Heckman CJ. Interactions between focused synaptic inputs and diffuse neuromodulation in the spinal cord. Ann N Y Acad Sci. 2010 Jun;1198:35-41. doi: 10.1111/j.1749-6632.2010.05430.x. PMID 20536918
- [Background] Heckman CJ, Mottram C, Quinlan K, Theiss R, Schuster J. Motoneuron excitability: the importance of neuromodulatory inputs. Clin Neurophysiol. 2009 Dec;120(12):2040-2054. doi: 10.1016/j.clinph.2009.08.009. Epub 2009 Sep 27. PMID 19783207
- [Background] Smulders K, Dale ML, Carlson-Kuhta P, Nutt JG, Horak FB. Pharmacological treatment in Parkinson's disease: Effects on gait. Parkinsonism Relat Disord. 2016 Oct;31:3-13. doi: 10.1016/j.parkreldis.2016.07.006. Epub 2016 Jul 17. PMID 27461783
- [Background] Kerr GK, Worringham CJ, Cole MH, Lacherez PF, Wood JM, Silburn PA. Predictors of future falls in Parkinson disease. Neurology. 2010 Jul 13;75(2):116-24. doi: 10.1212/WNL.0b013e3181e7b688. Epub 2010 Jun 23. PMID 20574039